CLINICAL TRIAL: NCT01211522
Title: MIND-USA Study: Modifying the Impact of ICU-Associated Neurological Dysfunction
Brief Title: The Modifying the Impact of ICU-Associated Neurological Dysfunction-USA (MIND-USA) Study
Acronym: MIND-USA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Wes Ely, Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG035117-01A1; 101082 (Other: Vanderbilt University Institutional Review Board)
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Delirium; Impaired Cognition; Long Term Psychologic Disorders
Keywords: Delirium; Intensive care; Mechanical ventilation; Antipsychotic; Haloperidol; Ziprasidone; Randomized; Placebo; Sepsis; Sedation; Long-term cognitive impairment
MeSH Terms: conditions — Delirium; Cognition Disorders; Sepsis | interventions — Haloperidol; ziprasidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind, placebo controlled
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Haloperidol (Experimental): Haloperidol
  Interventions: Drug: Haloperidol
- Ziprasidone (Experimental): Ziprasidone
  Interventions: Drug: Ziprasidone
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Haloperidol — Haloperidol, up to 10mg q12 hours, will be administered intravenously (IV) by bolus over up to 5 minutes at concentrations of 5mg/mL. Patient will only receive IV while in the ICU.
  Other Names: Haldol
  Arms: Haloperidol
Drug: Ziprasidone — Ziprasidone, up to 20mg q12 hours, will be administered intravenously (IV) by bolus over up to 5 minutes at concentrations of 10mg/mL. Patient will only receive IV while in the ICU.
  Other Names: Geodon
  Arms: Ziprasidone
Drug: Placebo — Placebo, up to 10mL q12 hours, will be administered intravenously (IV) by bolus over up to 5 minutes. Patient will only receive IV while in the ICU.
  Arms: Placebo

SUMMARY:
The long-term objective of the MIND-USA (Modifying the Impact of ICU-Induced Neurological Dysfunction-USA) Study is to define the role of antipsychotics in the management of delirium in vulnerable critically ill patients. We and others have shown that delirium is an independent predictor of more death, longer stay, higher cost, and long-term cognitive impairment often commensurate with moderate dementia. The rapidly expanding aging ICU population is especially vulnerable to develop delirium, with 7 of 10 medical and surgical ICU patients developing this organ dysfunction. Antipsychotics are the first-line pharmacological agents recommended to treat delirium, and over the past 30 years they gained widespread use in hospitalized patients globally prior to adequate testing of efficacy and safety for this indication. Haloperidol, the most commonly chosen antipsychotic, is used by over 80% of ICU doctors for delirium, while atypical antipsychotics are prescribed by 40%. Antipsychotics safety concerns include lethal cardiac arrhythmias, extrapyramidal symptoms, and the highly publicized increased mortality associated with their use in non-ICU geriatric populations. The overarching hypothesis is that administration of typical and atypical antipsychotics-haloperidol and ziprasidone, in this case-to critically ill patients with delirium will improve short- and long-term clinical outcomes, including days alive without acute brain dysfunction (referred to as delirium/coma-free days or DCFDs) over a 14-day period; 30-day, 90-day, and 1-year survival; ICU length of stay; incidence, severity, and/or duration of long-term neuropsychological dysfunction; and quality of life at 90-day and 1-year. To test these hypotheses, the MIND-USA Study will be a multi-center, double-blind, randomized, placebo-controlled investigation in 561 critically ill, delirious medical/surgical ICU patients who are (a) on mechanical ventilation or non-invasive positive pressure ventilation or (b) in shock on vasopressors. In each group (haloperidol, ziprasidone, and placebo), 187 patients will be enrolled and treated until delirium has resolved for 48 hours or to 14 days (whichever occurs first) and followed for 1 year.

DETAILED DESCRIPTION:
The primary and secondary outcomes of the MIND-USA investigation will be analyzed both according to the individual comparisons by group of "haloperidol treated" vs. "placebo treated" and "ziprasidone treated" vs. "placebo treated" and also the combined grouping of both antipsychotics ("haloperidol plus ziprasidone treated" patients vs. "placebo treated" patients). In the latter third of the study, as a result of a paper by Patel S et al AJRCCM 2014 about rapidly reversible delirium (RRD), we considered modifying delirium assessments to detect those who might convert from CAM-ICU positive to negative following SATs, but we estimated that only 5 patients per arm would be in this category (and indeed <20 per arm in the entire study using the 10% rate published by Patel). With such low numbers and the assurance that through randomization we would have all groups analyzed similarly according to the study drug assignment, we elected not to alter the protocol and not to conduct subgroup analyses according to RRD status.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients (≥18 years old)
2. in a medical and/or surgical ICU
3. on mechanical ventilation or non-invasive positive pressure ventilation (NIPPV), and/or requiring vasopressors due to shock
4. delirious (according to the CAM-ICU)

Exclusion Criteria:

1. Rapidly resolving organ failure criteria, indicated by planned immediate discontinuation of mechanical ventilation, NIPPV, and/or vasopressors at the time of screening for study enrollment
2. Pregnancy or breastfeeding (negative pregnancy test required prior to enrollment of female patients of childbearing age)
3. Severe dementia or neurodegenerative disease, defined as either impairment that prevents the patient from living independently at baseline or IQCODE >4.5, measured using a patient's qualified surrogate, mental illness requiring long-term institutionalization, acquired or congenital mental retardation, Parkinson's disease, Huntington's disease, and/or coma or another severe deficit due to structural brain disease such as stroke, intracranial hemorrhage, cranial trauma, intracranial malignancy, anoxic brain injury, or cerebral edema.
4. History of torsades de pointes, documented baseline QT prolongation (congenital long QT syndrome), or QTc >500 ms at screening due to refractory electrolyte abnormalities, other drugs, or thyroid disease
5. Ongoing maintenance therapy with typical or atypical antipsychotics
6. History of neuroleptic malignant syndrome (NMS), haloperidol allergy, or ziprasidone allergy
7. Expected death within 24 hours of enrollment or lack of commitment to aggressive treatment by family or the medical team (e.g., likely withdrawal of life support measures within 24 hours of screening)
8. Inability to obtain informed consent from an authorized representative within 72 hours of meeting all inclusion criteria, i.e., developing qualifying organ dysfunction criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2011-12-14 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2018-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Wesley Ely, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (16):
- United States (16):
  - Denver Health/University of Colorado Health Sciences Center, Denver, Colorado
  - Yale University Medical Center, New Haven, Connecticut
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Albert Einstein Medical College-Montefiore Medical Center, The Bronx, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Moses Cone Health System, Greensboro, North Carolina
  - The Ohio State Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Health Care System, Dallas, Texas
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Ahn S, LaNoue M, Su H, Moale AC, Scheunemann LP, Kiehl AL, Douglas IS, Exline MC, Gong MN, Khan BA, Owens RL, Pisani MA, Rock P, Jackson JC, Ely EW, Girard TD, Boehm LM. Post-Intensive Care Syndrome and Caregiver Burden: A Post Hoc Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2025 Apr 1;8(4):e253443. doi: 10.1001/jamanetworkopen.2025.3443. PMID 40198074
- [Derived] Mart MF, Boehm LM, Kiehl AL, Gong MN, Malhotra A, Owens RL, Khan BA, Pisani MA, Schmidt GA, Hite RD, Exline MC, Carson SS, Hough CL, Rock P, Douglas IS, Feinstein DJ, Hyzy RC, Schweickert WD, Bowton DL, Masica A, Orun OM, Raman R, Pun BT, Strength C, Rolfsen ML, Pandharipande PP, Brummel NE, Hughes CG, Patel MB, Stollings JL, Ely EW, Jackson JC, Girard TD. Long-term outcomes after treatment of delirium during critical illness with antipsychotics (MIND-USA): a randomised, placebo-controlled, phase 3 trial. Lancet Respir Med. 2024 Aug;12(8):599-607. doi: 10.1016/S2213-2600(24)00077-8. Epub 2024 Apr 30. PMID 38701817
- [Derived] Stollings JL, Boncyk CS, Birdrow CI, Chen W, Raman R, Gupta DK, Roden DM, Rivera EL, Maiga AW, Rakhit S, Pandharipande PP, Ely EW, Girard TD, Patel MB. Antipsychotics and the QTc Interval During Delirium in the Intensive Care Unit: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Jan 2;7(1):e2352034. doi: 10.1001/jamanetworkopen.2023.52034. PMID 38252439
- [Derived] Girard TD, Exline MC, Carson SS, Hough CL, Rock P, Gong MN, Douglas IS, Malhotra A, Owens RL, Feinstein DJ, Khan B, Pisani MA, Hyzy RC, Schmidt GA, Schweickert WD, Hite RD, Bowton DL, Masica AL, Thompson JL, Chandrasekhar R, Pun BT, Strength C, Boehm LM, Jackson JC, Pandharipande PP, Brummel NE, Hughes CG, Patel MB, Stollings JL, Bernard GR, Dittus RS, Ely EW; MIND-USA Investigators. Haloperidol and Ziprasidone for Treatment of Delirium in Critical Illness. N Engl J Med. 2018 Dec 27;379(26):2506-2516. doi: 10.1056/NEJMoa1808217. Epub 2018 Oct 22. PMID 30346242

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Haloperidol | Ziprasidone | Placebo
Started | 192 | 190 | 184
Completed | 189 | 183 | 179
Not Completed | 3 | 7 | 5
Not completed — Withdrawal by Subject | 3 | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Haloperidol | Ziprasidone | Placebo | Total
Number analyzed (Participants) | 192 | 190 | 184 | 566
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [51 to 69] | 61 [50 to 69] | 59 [52 to 67] | 60 [51 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 82 | 77 | 243
  Male | 108 | 108 | 107 | 323
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 23 | 27 | 26 | 76
  White | 163 | 151 | 153 | 467
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 12 | 5 | 23
Region of Enrollment [Number; unit: participants]
  United States | 192 | 190 | 184 | 566
Admission diagnosis [Count of Participants; unit: Participants]
  ARDS | 44 | 35 | 39 | 118
  Sepsis | 43 | 33 | 35 | 111
  Airway protection | 46 | 44 | 53 | 143
  COPD/asthma/other pulmonary | 20 | 28 | 23 | 71
  Surgery | 13 | 23 | 13 | 49
  CHF/MI/arrhythmia | 6 | 6 | 6 | 18
  Cirrhosis/liver failure | 3 | 3 | 6 | 12
  Seizures/neurologic disease | 4 | 1 | 1 | 6
  Other | 13 | 17 | 8 | 38

OUTCOME MEASURES:

1. Primary Outcome: Delirium/Coma-free Days (DCFDs)
Description: Defined as the number of days during the 14-day intervention period (beginning on the day of randomization) that the patient was alive and experienced neither delirium nor coma.
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Haloperidol | Ziprasidone | Placebo
Number analyzed (Participants) | 192 | 190 | 184
days | 8 [0 to 11] | 8 [2 to 11] | 7 [0 to 11]

2. Secondary Outcome: Mortality
Description: Deaths within the specified timeframe
Time Frame: 30-day and 90-day
Measure: Count of Participants; unit: Participants
Arm/Group | Haloperidol | Ziprasidone | Placebo
Number analyzed (Participants) | 192 | 190 | 184
Participants
  30-day mortality | 50 | 53 | 50
  90-day mortality | 73 | 65 | 63

3. Secondary Outcome: Delirium Duration
Description: Duration of delirium during the intervention period
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Haloperidol | Ziprasidone | Placebo
Number analyzed (Participants) | 192 | 190 | 184
days | 4 [2 to 7] | 4 [2 to 6] | 4 [2 to 8]

4. Secondary Outcome: Number of Participants With Torsades de Pointes
Time Frame: 14 days plus 4-day post-study drug period (if longer than 14 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Haloperidol | Ziprasidone | Placebo
Number analyzed (Participants) | 192 | 190 | 184
Participants | 2 | 0 | 0

5. Secondary Outcome: Number of Participants With Extrapyramidal Symptoms
Time Frame: 14 days plus 4-day post-study drug period (if longer than 14 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Haloperidol | Ziprasidone | Placebo
Number analyzed (Participants) | 192 | 190 | 184
Participants | 1 | 1 | 1

6. Secondary Outcome: Number of Participants With Neuroleptic Malignant Syndrome
Time Frame: 14 days plus 4-day post-study drug period (if longer than 14 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Haloperidol | Ziprasidone | Placebo
Number analyzed (Participants) | 192 | 190 | 184
Participants | 0 | 0 | 0

7. Secondary Outcome: Time to Liberation From Mechanical Ventilation
Description: Days from randomization to successful liberation from mechanical ventilation, where "successful" indicates that liberation was followed by at least 48 hours alive and without reinitiation of invasive or noninvasive ventilation.
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Haloperidol | Ziprasidone | Placebo
Number analyzed (Participants) | 192 | 190 | 184
days | 2 [1 to 6] | 3 [2 to 5] | 3 [1 to 5]

8. Secondary Outcome: Time to Final ICU Discharge
Description: Days from randomization to final, successful ICU discharge, where "successful" indicates that discharge was followed by at least 48 hours alive. "ICU discharge" is represented by readiness for ICU discharge indicated by a physician order for transfer to a lower level of care even if a bed availability problems prevent actual discharge from the ICU.
Time Frame: 90 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Haloperidol | Ziprasidone | Placebo
Number analyzed (Participants) | 192 | 190 | 184
days | 5 [3 to 13] | 6 [3 to 10] | 5 [3 to 14]

9. Secondary Outcome: Time to ICU Readmission
Description: Days from first ICU discharge to next ICU readmission.
Time Frame: 90 days after first ICU discharge
Population: Time to ICU readmission reported among those who were readmitted to the ICU
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Haloperidol | Ziprasidone | Placebo
Number analyzed (Participants) | 27 | 18 | 23
days | 5 [2 to 9] | 5 [2 to 9] | 4 [1 to 8]

10. Secondary Outcome: Time to Hospital Discharge
Description: Days from randomization to successful hospital discharge, where "successful" indicates that discharge was followed by at least 48 hours alive.
Time Frame: 90 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Haloperidol | Ziprasidone | Placebo
Number analyzed (Participants) | 192 | 190 | 184
days | 13 [8 to 22] | 12 [8 to 21] | 13 [8 to 23]

ADVERSE EVENTS:
Time Frame: During the period when the patients were receiving a trial drug or placebo and for 4 days after discontinuation, we assessed the patients for side effects. We also collected clinical outcomes data until hospital discharge or up to 90 days.
Arm/Group | Haloperidol | Ziprasidone | Placebo
All-Cause Mortality (participants affected / at risk) | 73/192 | 65/190 | 63/184
Serious Adverse Events (participants affected / at risk) | 3/192 | 1/190 | 1/184
Other Adverse Events (participants affected / at risk) | 55/192 | 70/190 | 56/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Haloperidol (N=192) | Ziprasidone (N=190) | Placebo (N=184)
Torsades de pointes (Cardiac disorders) | 2 | 1 | 1
Neuroleptic malignant syndrome (Nervous system disorders) | 0 | 0 | 0
Extrapyramidal symptoms (Nervous system disorders) | 1 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Haloperidol (N=192) | Ziprasidone (N=190) | Placebo (N=184)
Oversedation (Nervous system disorders) | 42 | 50 | 46
Prolonged QTc (Cardiac disorders) | 13 | 20 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-06-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT01211522/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT01211522/SAP_001.pdf